CLINICAL TRIAL: NCT02622347
Title: Spiking-and-Recovery Experiment DOREMI Study
Status: Completed | Type: Observational
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Bart CJM Fauser, prof. dr. F.J.M. Broekmans, UMC Utrecht
Other Study IDs: rFSH Spiking Experiment
Record Dates: First submitted 2015-12-02; First posted 2015-12-04 (Estimated); Last update posted 2017-05-16 (Actual); Status verified 2017-05

CONDITIONS: FSH Assay

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — Bloodserum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to test the validity of our in-house chemiluminescence assay for measurement of folliclestimulating hormone (FSH) serum levels before and during exogenous recombinant FSH (rFSH) administration.

DETAILED DESCRIPTION:
Study question Does our in-house Beckman-Coulter Unicel DXi800 (Woerden, the Netherlands) chemiluminescence assay completely and consistently recover added known quantities of FSH on top of a known basal serum FSH concentration?

Spiking-recovery experiment The investigators propose a spiking-recovery experiment in which 30 serum samples of different women with basal FSH concentration varying between 0-14 IU/L will be divided into two equal volume parts and spiked with a specific concentration of rFSH (Gonal-F, follitropin alpha; Merck Serono) which will provide a calculated rise in FSH concentration similar to in vivo serum levels.

To perform more reliable testing, the samples will be tested over multiple days.

Basal FSH spiking experiment In the table below an example is given of different basal FSH levels spiked with rFSH diluted 2000 times and the theoretical rise in serum that should be established.

Gonal F concentration is 600 U/L but this concentration unit cannot directly be compared to the units used for the for the routine serum FSH measurement (IU/L). From a pilot experiment the investigators know that on average 60% of rFSH is picked up by the Beckman-Coulter assay.

Buffer spiking In order to determine whether recovery is also influenced by properties of blood serum, the investigators will conduct another spiking experiment in which different concentrations of rFSH will be added to an amount of buffer, with no basal [FSH]; 0,1 M phosphate buffer, pH 7.4 with 1-2% of bovine serum albumin (BSA). A calibration line will be constructed with 6 concentrations of recF: range 0-40 U/L.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Basal FSH concentration varying between 0-14 IU/L

Exclusion Criteria:

* None

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Bloodserum samples of 30 women with basal FSH concentration varying between 0-14 IU/L.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-08; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Recovery rate | 1 day
  Recovery rate of recombinant FSH in blood serum as measured by our in-house assay

CONTACTS AND LOCATIONS:
Overall Officials: Broekmans, Principal Investigator — UMC Utrecht
Locations (1):
- UMC Utrecht, Utrecht, Netherlands